CLINICAL TRIAL: NCT06211686
Title: The Effectiveness of a Health Promotion Program for Older People With Post-Covid-19 Sarcopenia
Acronym: Sarcopenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mahidol University (Other)
Collaborators: National Health Security Office, Thailand (Other)
Responsible Party: Principal Investigator, Wanabhorn Tongchom, Principle investigator, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MURA2023/918; 2023/918 (Other: MURA)
Record Dates: First submitted 2023-12-28; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Post COVID-19 Condition
Keywords: Sarcopenia; Older people; Health Promotion Program; Post COVID-19
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: Phase I: Descriptive survey research Phase II: Quasi-experimental research
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Protein supplement and Resistance exercise (Experimental)
  Interventions: Other: Protein powder and Resistance exercise

INTERVENTIONS:
Other: Protein powder and Resistance exercise — 1. Protein powder supplementation 25-30 g/day
  2. Resistance exercise 2 time/week

SUMMARY:
The goal of this clinical trial is to investigate the prevalence of sarcopenia in older people with post-COVID-19 living in Ratchatewi district, Bangkok and to test the effectiveness of health promotion program for older people with post-COVID-19 Sarcopenia. The main questions it aim to answer are: • How many is the prevalence of sarcopenia in older people with post-COVID-19 living in Ratchatewi district, Bangkok? • Can the health promotion program improve muscle mass and muscle strength in older people with post-COVID-19 Sarcopenia ? Participants will be asked eating protein supplement one scoop /day and exercising 2 times/week for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Older people with post-COVID-19 sarcopenia aged more than and equal 60 years
* No disabilities
* Able to read, write and communicate Thai langue
* Live in Bangkok
* Moderate post-covid-19 state defined by Thai version of the COVID-19 Yorkshire Rehabilitation Scale
* No soy protein allergy
* Sign inform consent

Exclusion Criteria:

* Severe post-covid-19 state defined by Thai version of the COVID-19 Yorkshire Rehabilitation Scale and complicated health problems
* Disabilities
* Unable to read, write and communicate Thai langue
* Soy protein allergy
* CKD 4 and CKD 5
* Deny or withdraw from project

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Muscle mass | 3 months
  Muscle mass will be measured using BIA and calf circumference in kilograms.
Muscle strength | 3 motnhs
  Muscle strength will be assessed using hand grip strength in kilograms.
Physical fitness | 3 months
  Physical fitness will be measured using the Five Times Sit to Stand Test (FTSST) in second.

SECONDARY OUTCOMES:
Prevalence of sarcopenia | 3 months

IPD SHARING:
Plan to Share IPD: No